CLINICAL TRIAL: NCT04018391
Title: The TENDAI Study: Task Shifting to Treat Depression and HIV Medication Nonadherence in Low Resource Settings
Brief Title: Task Shifting to Treat Depression and HIV Medication Nonadherence in Low Resource Settings
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Massachusetts General Hospital (Other); University of Zimbabwe College of Health Sciences (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr Melanie Abas, Associate Professor in Global Mental Health, King's College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRCZ/A/2390; 1R01MH114708-01A1 (NIH)
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections; Depression
Keywords: HIV treatment; Depression; Medication Adherence
MeSH Terms: conditions — HIV Infections; Depression; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped care for non-adherence and depression (Experimental): Participants will be randomized approximately two weeks post-baseline. Those randomized to the experimental condition will receive the Intervention and Stepped Care Treatment Protocol
  Interventions: Behavioral: Stepped care for nonadherence and depression
- Enhanced Usual Care (Active Comparator): Participants will be randomized two weeks post-baseline. Those randomized to the control condition will receive Enhanced Usual Care.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Stepped care for nonadherence and depression — * Problem Solving for Depression and Adherence: A 6-session adherence and depression intervention based on a culturally adapted LifeSteps and Problem Solving Therapy for Depression.
  * Stepped Care Assessment for Antidepressant Treatment: If a participant's depression score remains above threshold in Session 6, the study interventionist will refer the participant to a Research Mental Health Nurse for a psychopharmacological assessment to prescribe an antidepressant to augment Problem Solving for Depression and Adherence.
  Arms: Stepped care for non-adherence and depression
Other: Enhanced Usual Care — Enhanced Usual Care: A combination of 1) clinic-provided adherence counseling, 2) access to providers trained in the World Health Organization Mental Health Gap Intervention Guide (mhGAP), 3) a letter to the participant's medical provider detailing the depression diagnosis, 4) access to the treatment components of the TENDAI intervention at no cost, after the participant has completed their 12-month follow-up assessment.
  Arms: Enhanced Usual Care

SUMMARY:
A hybrid effectiveness-efficacy trial to evaluate a stepped care task shifted intervention to treat depression and HIV medication nonadherence in low resource settings in rural Zimbabwe.

DETAILED DESCRIPTION:
Depression is commonly co-morbid with HIV infection in Zimbabwe and is consistently associated with worse adherence to antiretroviral therapy (ART). A task-shifted intervention for depression and ART adherence, suitable for delivery by non-specialists, could make a critical difference to the health and survival of people managing the challenges of HIV treatment in Zimbabwe. The TENDAI trial is a two-arm randomized controlled trial of an intervention for people on ART with viral non-suppression and clinically significant depression. It will be delivered at an HIV clinic in Marondera. TENDAI is a collaboration between the Department of Psychiatry, University of Zimbabwe College of Health Sciences, King's College London Institute of Psychiatry, Psychology and Neuroscience (London UK), and the Department of Psychiatry at Massachusetts General Hospital / Harvard Medical School.

ELIGIBILITY:
Inclusion Criteria:

* Initiated on ART for at least 6 months
* Clinically significant depression symptoms scoring >/= 10 on the Patient Health Questionnaire-9
* Viral non-suppression in past two months per local clinic standard (VL > 1000 copies/mL)
* Able to provide informed consent
* If prescribed antidepressants, on stable regimen for at least 2 months

Exclusion Criteria:

* Unable to provide informed consent
* Active major mental illness (e.g. untreated psychosis or mania, actively suicidal), major untreated or undertreated mental illness or advanced physical disease or severe cognitive impairment assessed using the psychosis module of the MINI, the PHQ-9, and the International HIV dementia Scale which would interfere with engagement in PST-AD
* Has ever received PST or CBT for depression
* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression | 12 - month post randomization study visit
  Viral Suppression operationalized as proportion of participants who achieve viral suppression (<1000 copies/mL)

SECONDARY OUTCOMES:
Depression severity | 12-month post randomization study visit
  Depression at 12 months post randomization measured as the total score on the Patient Health Questionnaire (PHQ-9). Each of the nine items is scored from 0 (not at all) to 3 (nearly every day). It is used as a continuous score ranging from 0 (no depressive symptoms) to 27 (all symptoms occurring daily/nearly daily).
Adherence to ART medication | 4 month post randomization study visit
  Adherence to ART medication, assessed as proportion of the sample achieving at least 90% adherence in the past month via pharmacy refill data
Adherence to ART medication | 12 month post randomization study visit
  Adherence to ART medication, assessed as proportion of the sample achieving at least 90% adherence in the past month via pharmacy refill data
Adherence to ART medication | 8 month post randomization study visit
  Adherence to ART medication, assessed as proportion of the sample achieving at least 90% adherence in the past month via pharmacy refill data
Self-reported adherence to ART medication | 4 month post randomization study visit
  Self-reported adherence to ART medication, assessed as the frequency of adherence in the past 30 days
Self-reported adherence to ART medication | 12 month post randomization study visit
  Self-reported adherence to ART medication, assessed as the frequency of adherence in the past 30 days
Self-reported adherence to ART medication | 8 month post randomization study visit
  Self-reported adherence to ART medication, assessed as the frequency of adherence in the past 30 days
Viral load copies/mL | 12-month post randomization study visit
  Viral load copies/mL assessed via Mean Log Viral Load

OTHER OUTCOMES:
Cost effectiveness of TENDAI Intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Melanie Abas, Principal Investigator — King's College London
Locations (1):
- Marondera Provincial Hospital, Marondera, Mashonaland East Province, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abas M, Mangezi W, Nyamayaro P, Jopling R, Bere T, McKetchnie SM, Goldsmith K, Fitch C, Saruchera E, Muronzie T, Gudyanga D, Barrett BM, Chibanda D, Hakim J, Safren SA, O'Cleirigh C. Task-sharing with lay counsellors to deliver a stepped care intervention to improve depression, antiretroviral therapy adherence and viral suppression in people living with HIV: a study protocol for the TENDAI randomised controlled trial. BMJ Open. 2022 Dec 5;12(12):e057844. doi: 10.1136/bmjopen-2021-057844. PMID 36576191